CLINICAL TRIAL: NCT04976218
Title: Phase Ⅰ Study of EGFR Targeted TGFβR-KO CAR T Cells in the Treatment of Previously Treated Advanced EGFR-positive Solid Tumors
Brief Title: TGFβR-KO CAR-EGFR T Cells in Previously Treated Advanced EGFR-positive Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Bio-therapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-067
Record Dates: First submitted 2021-07-19; First posted 2021-07-26 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Solid Tumor, Adult; EGFR Overexpression

STUDY DESIGN:
Intervention Model Description: TGFβR-KO CAR-EGFR T Cells will be administered to eligible patients in a 3+3 dose escalation manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Enrolled patients in this arm will be administered TGFβR-KO CAR-EGFR T Cells in 3+3 based escalation manner.
  Interventions: Biological: TGFβR-KO CAR-EGFR T Cells

INTERVENTIONS:
Biological: TGFβR-KO CAR-EGFR T Cells — Enrolled patients will be administered TGFβR-KO CAR-EGFR T Cells in 3+3 based escalation manner. The infused CAR+ T cell dose in phase IA will be started initially at 1-2×10^5/kg, dose 2 will be 1×10^6/kg，and dose 3 will be 1×10^7/kg, if DLT occurs in dose level 3, the following dose will return to 5×10^6/kg. In expansion period, the dose of infused CAR+ T cells will be determined by the recommended cell dose from phase IA.

SUMMARY:
Chimeric antigen receptor modified T (CART) cell therapy has been identified as a breakthrough therapy in hematologic malignancies. However, CART cell therapy yielded no satisfactory efficacy data in the study of solid tumors. One of major challenges is the complicated immunosuppressive tumor microenvironment (TME) in solid tumors. It has been reported that transforming growth factor-β (TGF-β) is one of the major regulatory factors in the TME. In this study, we construct CAR-EGFR-TGFβR-KO T cell by knocking out TGF-β receptor Ⅱ through CRISPR/Cas9 in order to study the anti-tumor activities and safety profiles of CAR-EGFR-TGFβR-KO T cell in previously treated advanced EGFR positive solid tumors.

DETAILED DESCRIPTION:
Chimeric antigen receptor modified T (CART) cell therapy has been identified as a breakthrough therapy in hematologic malignancies. Different from the promising efficacy in leukemia, lymphoma and multiple myeloma, however, CART cell therapy yielded no satisfactory efficacy data in the study of solid tumors. One of major challenges is the complicated immunosuppressive tumor microenvironment (TME) in solid tumors. It has been reported that transforming growth factor-β (TGF-β) is one of the major regulatory factors in the TME, which plays a key role in promoting tumor initiation, metastasis, and suppressing anti-tumor immunity. In this phase Ⅰstudy, we plan to construct CAR-EGFR-TGFβR-KO T cell by knocking out TGF-β receptor Ⅱ through CRISPR/Cas9 in order to study the anti-tumor activities and safety profiles of CAR-EGFR-TGFβR-KO T cell in the treatment of previously treated advanced EGFR antigen overexpressing solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years with estimated life expectancy >3 months.
2. Histopathological confirmed advanced solid tumors failed to at least first-line standard treatment. EGFR antigen expression level ≥ 50%.
3. Have at least one measurable target lesion.
4. Fresh solid tumor samples or formalin-fixed paraffin embedded tumor archival samples within 6 months are necessary; Fresh tumor samples are preferred. Subjects are willing to accept tumor re-biopsy in the process of this study.
5. Previous treatment must be completed for more than 4 weeks prior to the enrollment of this study, and subjects have recovered to <= grade 1 toxicity.
6. Have an Eastern Cooperative Oncology Group performance status (ECOG) of 0 or 2 at the time of enrollment.
7. Have adequate organ function, which should be confirmed within 2 weeks prior to the first dose of study drugs.
8. Previous treatment with anti-PD-1/PD-L1 antibodies are allowed.
9. Ability to understand and sign a written informed consent document.
10. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and up to 90 days after the last dose of the drug.

Exclusion Criteria:

1. Active, known or suspected autoimmune diseases.
2. Known brain metastases or active central nervous system (CNS). Subjects with CNS metastases who were treated with radiotherapy for at least 3 months prior to enrollment, have no central nervous symptoms and are off corticosteroids, are eligible for enrollment, but require a brain MRI screening.
3. Subjects are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
4. History of severe hypersensitive reactions to other monoclonal antibodies.
5. History of allergy or intolerance to study drug components.
6. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
7. History or concurrent condition of interstitial lung disease of any grade or severely impaired pulmonary function.
8. Uncontrolled intercurrent illness, including ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations and any other illness that would limit compliance with study requirements and jeopardize the safety of the patient.
9. History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
10. Pregnant or breast-feeding. Women of childbearing potential must have a pregnancy test performed within 7 days before the enrollment, and a negative result must be documented.
11. Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
12. Vaccination within 30 days of study enrollment.
13. Active bleeding or known hemorrhagic tendency.
14. Subjects with unhealed surgical wounds for more than 30 days.
15. Being participating any other trials or withdraw within 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects occuring treatment related adverse events | Up to 24 weeks following the infusion of TGFβR-KO CAR-EGFR T cells.
  Determining the safety profile following the initiation of treatment and grading these toxicities by CTCAE v5.0

SECONDARY OUTCOMES:
The percentage of enrolled patients that respond to TGFβR-KO CAR-EGFR T cell therapy. | Up to 24 weeks following the infusion of TGFβR-KO CAR-EGFR T cells.
  Overall response rate is defined as the sum of partial responses and complete responses
The percentage of enrolled patients alive and without progression at 6 months | 6 months
  Progression free survival (PFS) is defined as the time from enrollment to documented disease progression or death. Progression will be defined clinically or on imaging as per immune related response evaluation criteria in solid tumors (irRECIST) definition.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, PhD, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China